CLINICAL TRIAL: NCT02539043
Title: Effects of Ultrasound Cavitation Focused on Located Adiposity: Pilot Study
Brief Title: Effects of Ultrasound Cavitation Focused on Located Adiposity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Patricia Viana da Rosa, Adjunct Professor, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36341214.3.00005345
Record Dates: First submitted 2015-07-13; First posted 2015-09-02 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-08

CONDITIONS: Subcutaneous Fat
Keywords: Lipolysis; Subcutaneous Fat, Abdominal/metabolism; Subcutaneous Fat, Abdominal/ultrasonography; High-Intensity Focused Ultrasound Ablation/methods; Waist Circumference; Pilot Projects; Subcutaneous Fat; High-Intensity Focused Ultrasound Ablation; Adiposity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Focused ultrasound cavitation: Lipofocus (Active Comparator): The first group will receive only the application of focused ultrasound cavitation.
  Interventions: Device: LIPOFOCUS
- Focused ultrasound and drainage: Lipofocus (Active Comparator): The second group will receive focused ultrasound cavitation followed by stereodynamic drainage.
  Interventions: Device: LIPOFOCUS

INTERVENTIONS:
Device: LIPOFOCUS — In cavitation focused ultrasound procedure for reduction of localized abdominal fat, the parameters will be used: maximum power of 8 Watts at a frequency of 1 Megahertz (MHz), and the transducer is used in a timely manner by performing a sweep of the area by 03 times, at random.
  Arms: Focused ultrasound cavitation: Lipofocus
Device: LIPOFOCUS — In cavitation focused ultrasound procedure for reduction of localized abdominal fat, the parameters will be used: maximum power of 8 Watts at a frequency of 1 MHz, and the transducer is used in a timely manner by performing a sweep of the area by 03 times, at random . The procedure is followed by stereodynamic drainage, where it will be used a printhead comprising three ERAs (effective radiation area) of 15 Watt each time this procedure is calculated through the area (size of the area to be treated) divided by ERA (cm² head size).
  Arms: Focused ultrasound and drainage: Lipofocus

SUMMARY:
The aim of this study is to evaluate the effect of cavitation ultrasound focused on localized adiposity and its effects associated with stereodynamic lymphatic drainage. The investigators aim also to know if this procedure will influence the biochemical profile of the individuals concerned, as well as whether it will be found difference between the group that will receive focused ultrasound cavitation associated with stereodynamic drainage and the group will receive only focused cavitation ultrasound.

DETAILED DESCRIPTION:
This study will be a double-blind randomized clinical trial, preceded by a pilot study due to lack of data in the literature impossible to calculate the size of adequate sample.

The overall objective of the study is to evaluate the effect of cavitation ultrasound focadalizado in localized adiposity and its associated lymphatic drainage effects stereodynamic.

The specific objectives are:

Evaluate and compare the effects of focused ultrasound cavitation in reducing hypodermic layer and anthropometric measurements of women; To evaluate the acute and chronic effects of the technique; To evaluate the reduction in adipose tissue layer from the ultrasound image; Evaluate and compare the reduction of the fat layer through intergroup and intragroup photographic image; Evaluating and comparing serum biochemical parameters (total cholesterol, triglycerides, HDL cholesterol, LDL cholesterol, glucose, urea and creatinine) of women undergoing focused ultrasound cavitation; Evaluate and compare the technical efficiency in group A (without stereodynamic drainage) and B (with stereodynamic drainage).

This study will be conducted with 28 volunteers, respecting the criteria for inclusion and exclusion previously cited by reading and signing of the free and clear consent. Participants will be divided into 02 groups randomly. Randomization will be performed by using the local random distribution www.random.org tool, in order to prevent the researcher to identify which intervention will be performed on each patient. The generation of sequence numbers shall be made by the researcher "blind" to the study, after the selection of patients for inclusion and exclusion criteria. The sequence numbers to be used for randomization will be kept confidential until such time as the intervention Participants will undergo a 4-week control period between the first (base) and the second evaluation (pre-treatment), so each participant It will be their own control, ensuring that the possible changes that may be found at the end of the project will be related to the procedure and not influenced by lifestyle habits. During the period the research subjects will be instructed not alterararem their respective routine activities.

08 sessions will be conducted Cavitational Focused Ultrasound in individual applications, once per week, total of 08 weeks of treatment. The first collection (pre-treatment) will be only to carry out the data collection.

Data collection will consist of:

* Questionnaire of habitual physical activity Baecke - in the base period will be asked participants to answer this quiz to knowledge of their routine physical activity;
* Perimetry - anthropometric measurements will be measured by a previously trained evaluator. During the measurement of the circumference of the tape will be adjusted to the body, directly on the skin in order to provide more reliable measurements possible, without the occurrence of tape pressure on subcutaneous tissue causing deformity. These data will be verified in four stages: pre-treatment, before the first session after the first session and after the eighth treatment session. They will be measured:

Height: will be determined by the balance rule coupled with a degree in 1 mm, with the individual back to this, in an upright standing position, feet together, and trying to put the posterior surface of heels, pelvic and shoulder girdle contact instrument; Body weight will be measured through traditional mechanical scale with 100g graduation, with front man for the same, in the upright position, feet together, wearing light clothes and without shoes; Body Mass Index (BMI) - Based on height and weight will be held calculate BMI, kg ÷ height x height; Abdominal skin fold, used to estimate the percentage of body fat will be taken using caliper. It will be measured abdominal crease, having as anatomical reference umbilicus, plying up the region located 1 to 3 cm to the right of scar parallel to the longitudinal axis of the body; Waist circumference will be measured using the measuring tape positioned parallel to the ground, where the measurement is taken over previous iliac crests 5 cm above the previous iliac crests 10 cm above the iliac crest and waist earlier; Hip circumference, the tape measure is parallel to the ground and positioned in terms of points of trocantéricos right and left, while the individual will be assessed with feet together; Thigh circumference will also feature the same principles described above, but will be used as an indication of circumference changes that are unrelated to treatment, such as changes induced by weight loss.

* Bioimpedance - Evaluations shall be performed by a professional with training and experience in this type of analysis. Obtaining the bioimpedance will take place in two stages: in the base period (pre-treatment) and after the end of treatment (after the eighth session). For the examination, it will be used Maltron BF-900 model system and will be adopted the protocol recommendations proposed by the European Society for Clinical Nutrition and Metabolism: To assess body mass and height of the individual at the time of examination; Fasting individual and not drink alcohol for at least 8 hours; Urinate before the exam; Not perform physical exercise in the eight hours before the test; No injury to the skin where the electrode will be; Clean the skin with alcohol; Position the electrodes always on the same side of the body; Minimum 5 cm distance between the electrodes; Separate arms of the trunk for 30 ° and 45 ° legs apart; The environment duty will be neutral (no electric or magnetic field); It should be observed body shape for the risk of any possible anomaly (edema, amputation, atrophy, scoliosis, dystrophy); When prostheses or implants, is measured on the opposite side (KYLE et al, 2004); You can not use metal objects during the examination as earrings, bracelets, watches and the like; There may be conducted in subjects who have pacemaker and who are in pregnancy.
* Ultrasound diagnosis - will be used to analyze and measure the hypodermic layer of the assessed region. This will be measured by a professional with training and experience in this type of evaluation. The evaluator will collect the images in the basic period (4 weeks before the start of treatment) before the first and after the last login session. The results will be examined by a software in order to assess the thickness and statistics of the images defined by the image of ultrasound. To collect the individual will be in the supine position, the head is positioned above the navel and the fat thickness is measured from the inner layer of the skin to the aponeurosis of the rectus abdominis muscle in the middle of the Alba line area. The fat thickness measurement is performed with linear probe (7.5 MHz) with a depth of 4 to 5 cm.
* Blood collection - The analyzes will be performed on serum obtained by venipuncture, after an overnight fast of 12 hours. 02 will be held series of biochemical assessment by patient, where each collection will last for a maximum of 30 seconds. The first sample time is performed at baseline, i.e., before the control period. The second collection will be held after the end of treatment Focused Ultrasound Cavitational. After harvesting, the material is centrifuged at 3500 rpm / 10 minutes and then the analysis will be performed. Samples will be collected by a person trained for this, with latex glove use. They will be analyzed: total cholesterol, triglycerides, HDL cholesterol, LDL cholesterol, glucose, urea and creatinine.
* Photo documentation - To carry out the photos, there will be a standard procedure in order to maintain quality, the angle and the light always the same, so that the observed results can be compared reliably. Initially, patients using swimsuits, will be photographed standing in front and lateral planes (both sides) parallel to the plane of the camera sensor. The camera is mounted on the tripod, level and horizontal position, with the 105mm lens will be placed in proper height for framing the abdominal region, and at a distance of 1 meter. The flash is mounted on the hot shoe of the camera, set in TTL mode with the driven diffuser and will have its head directed forward. The camera will be displayed in manual mode, with f5.6 aperture, shutter speed to 1/60 second and ISO 200. The images will be taken in the base period and after the treatment and will be recorded in RAW format. The computational treatments on the images will be made in batch, so that all images suffer the same treatment and will be transformed into shades of gray. For image analysis, randomization of the resulting photographs will be held, and they will be delivered to two blind evaluators (physiotherapists) who will be invited to participate in the project to carry out this analysis. They will not know which patient images belong, or what the correct order of application of images. The evaluation will be as follows: both receive the photos in random order and will have to put them in progression order of the sessions, in 2 times: before and after treatment. After the correct organization, assess images qualitatively. Importantly, the designated evaluator will be a person with extensive knowledge about the procedure. The photographic analysis will be performed in two stages:

Step 1: The evaluators will receive slides with 6 photos for each patient, in random order (will be photographs in black and white, not to interfere in the result). The evaluator will classify the images in the order of 1 to 2, being 1 before treatment, after treatment and 2 referring to the reduction of localized fat deposits in the abdominal region (it is expected that the treatment reduces the action of the abdominal region, so this sort order). They will receive 3 slides for each patient, each containing images of the respective regions measured: front, right profile and left profile.

Step 2: evaluators should classify the changes in the abdominal region, in one of the degrees of the scale below: 0% = no change; 1% - 25% = little change; 25-50% = was no change in terms of improvement, but nothing extremely significant; 50% or more = a change from the reduction of localized fat in the abdominal area is visible / improved considerably.

ELIGIBILITY:
Inclusion criteria:

* Females, showing adiposity located in the abdominal area;
* Body Mass Index values are within normal values, 18.5 kg / m2 and 24.9 kg / m2;
* Patients must agree and sign the consent form and clarified.

Exclusion criteria:

* Individuals who contraceptive hormone therapy was changed for less than 4 weeks of starting treatment;
* Showing as lower skinfold to 2 cm;
* Making use of anti-dyslipidemic drugs;
* Present areas of hypoesthesia at the injection site;
* Having inflammation or infection in the region to be treated;
* Woman in pregnancy or breastfeeding;
* With clinical history of malignancies;
* Who have metal implants or cardiac pacemaker;
* Presenting coagulation disorders or making use of medications that alter blood clotting;
* Patients with osteoporosis and / or diabetes mellitus.

Ages: 19 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2015-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Use of Ultrasound Focused Cavitational reduce the layer of fat in the abdominal area abdominal region. | Eight weeks
Use of Ultrasound Focused Cavitational associated with stereodynamic drainage reduce the layer of fat in the abdominal region. | Eight weeks

CONTACTS AND LOCATIONS:
Overall Officials: Cinara LS Lima, Principal Investigator — Federal University of Health Science of Porto Alegre; Suélen A Kislowski, Principal Investigator — Federal University of Health Science of Porto Alegre